CLINICAL TRIAL: NCT00749281
Title: Neutrophil Gelatinase-associated Disease: a Potential Biomarker of the Severity of Coronary Artery Disease
Brief Title: Neutrophil Gelatinase-associated Lipocalin Concentration in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Cardiovascular Research Society, Greece (Other)
Responsible Party: Department of Cardiology, Athens Euroclinic
Other Study IDs: 3.8.9.2008
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: atherosclerosis; ngal; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with angiographically confirmed significant CAD
- 2: Patients without significant CAD

SUMMARY:
Serum NGAL has been described as a biomarker of neutrophil activation and an inflammatory marker which correlates to obesity and its metabolic complications. Since neutrophil activation has been implicated in the pathogenesis of coronary artery disease, the investigators hypothesized that serum NGAL levels would be higher in patients with CAD and that serum concentration would correlate with the extent of CAD as documented by coronary angiography, serving as a potential biomarker of the severity of CAD.

DETAILED DESCRIPTION:
Inflammation is considered to play a major role in coronary artery disease (CAD) which accounts for high morbidity and mortality rates in the western world. Several lines of evidence support a role for neutrophils in the development of atherosclerosis and its progression.

Neutrophil gelatinase-associated lipocalin (NGAL), also known as Lipocalin-2, is a 25-kDa secretory glycoprotein that was originally identified in mouse kidney cells and human neutrophil granules. This protein has been used as a marker of neutrophil activation in several studies, while recently it was found to be an inflammatory marker closely related to obesity and its metabolic complications.

Recently, lactoferrin, a protein which co-localizes with NGAL in the specific granules of human neutrophils has been proposed as a more dynamic marker of neutrophil activation compared to the widely used myeloperoxidase in patients with CAD.

In line with the accumulating evidence, this study is designed to investigate the relationship between serum NGAL concentration and the presence or the severity of coronary artery disease according to coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients undergoing coronary angiography due to suspected CAD based on clinical history and results from non-invasive testing

Exclusion Criteria:

* Abnormal renal function
* Any known active inflammatory disease
* Receiving medical therapy with antibiotics, corticosteroids, immunosuppressive agents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demosthenes Katritsis, MD,PhD, Study Chair — Athens Euroclinic and Cardiovascular Research Society
Locations (1):
- Athens Euroclinic, Athens, Attica, Greece